CLINICAL TRIAL: NCT02942524
Title: Tool to Engage Patients in Discharge (TEPID)
Brief Title: Checklist Tool in Engaging Patients in the Discharge Planning Process
Acronym: TEPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Lisa Graham, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-14237; NCI-2016-01308 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-10-21; First posted 2016-10-24 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Hospitalization; Malignant Neoplasm; Transitional Care Planning
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (TEPID) (Experimental): Patients complete the TEPID checklist of items during hospital stay.
  Interventions: Other: Communication Intervention; Other: Questionnaire Administration; Other: Survey Administration

INTERVENTIONS:
Other: Communication Intervention — Complete TEPID
Other: Questionnaire Administration — Ancillary studies
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well a checklist tool works in engaging patients in the discharge planning process. Engaging patients in the discharge process may increase participation in the discharge process and improve discharge outcomes, understanding of care after hospitalization, and decrease complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Measure the impact on discharge and transition satisfaction of utilizing questions from the Consumer Assessment of Healthcare Providers and Systems (CHAPS) patient satisfaction survey.

II. Measure the impact of the Tool to Engage Patients in Discharge (TEPID) on patient's Readiness for Hospital Discharge and Problems After Discharge Questionnaire-English (PADQ-E) results.

III. Measure the impact on decreasing healthcare utilization measures: readmission rates within 30 days from hospital discharge, hospital length of stay of admission in hospital, and emergency department visits within 30 days of hospital discharge.

OUTLINE:

Patients complete the TEPID checklist of items during hospital stay.

After completion of the study, patients are followed up for 35 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients fluent in English, conscious, coherent, and alert or have an adult caregiver present that is fluent in English will be identified for the TEPID research project

Exclusion Criteria:

* Patients discharged to another inpatient facility (hospice, skilled nursing facility, long term acute care hospital [LTACH], or acute rehab) or patients discharged home with hospice will be excluded
* Any patients that are transferred to another unit prior to discharge will be excluded

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-04 (Actual)

PRIMARY OUTCOMES:
Average score from the PADQ-E | Up to 12 months
  A simple analysis of variance (ANOVA) model with floor as a fixed blocking factor treatment (TEPID or no TEPID) as a fixed factor. Unit appears in the model as a nested factor within treatment, and statistical tests will be adjusted for this nesting structure. The main test of interest in each model is the overall effect of treatment, which quantifies the effect of TEPID on the average score for the response. P-values below 0.05 for this effect will be considered statistically significant.
Average score from the Readiness for Hospital Discharge Scale | Up to 12 months
  A simple ANOVA model with floor as a fixed blocking factor treatment (TEPID or no TEPID) as a fixed factor. Unit appears in the model as a nested factor within treatment, and statistical tests will be adjusted for this nesting structure. The main test of interest in each model is the overall effect of treatment, which quantifies the effect of TEPID on the average score for the response. P-values below 0.05 for this effect will be considered statistically significant.
Emergency department visits | Up to 12 months
  A generalized linear model will be used for the binary responses (readmission and ED visit).
Patient satisfaction as measured by the Press Ganey Consumer Assessment of Healthcare Providers and Systems Survey | Up to 12 months
  A simple ANOVA model with floor as a fixed blocking factor treatment (TEPID or no TEPID) as a fixed factor. Unit appears in the model as a nested factor within treatment, and statistical tests will be adjusted for this nesting structure. The main test of interest in each model is the overall effect of treatment, which quantifies the effect of TEPID on the average score for the response. P-values below 0.05 for this effect will be considered statistically significant.
Readmission rates | Up to 12 months
  A generalized linear model will be used for the binary responses (readmission and ED visit).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Graham, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: jamesline — http://cancer.osu.edu